CLINICAL TRIAL: NCT01235065
Title: GlideScope vs. Direct Laryngoscope for Emergency Intubation
Brief Title: GlideScope Versus Direct Laryngoscope for Emergency Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HP-00042451
Record Dates: First submitted 2010-10-22; First posted 2010-11-05 (Estimated); Results first posted 2023-06-01 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2018-06

CONDITIONS: Oral Intubation
Keywords: airway management; trauma; intubation
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- direct laryngoscope (Active Comparator): emergency intubation with direct laryngoscopy technique
  Interventions: Device: type of laryngoscope
- video laryngoscope (Active Comparator): emergency intubation with video laryngoscopy technique
  Interventions: Device: type of laryngoscope

INTERVENTIONS:
Device: type of laryngoscope — Patients who require emergency rapid sequence intubation are randomized to intubation with either the direct laryngoscope or the video laryngoscope
  Other Names: Macintosh direct laryngoscope vs. GlideScope video laryngoscope

SUMMARY:
The purpose of this study is to assess if the GlideScope video laryngoscope is superior to the Macintosh direct laryngoscope for definitive airway management in acutely-injured patients.

DETAILED DESCRIPTION:
On admission to the emergency department following traumatic injury, many patients require placement of an artificial airway to support their breathing, provide oxygen and protect their airway. This procedure is accomplished through a number of different techniques and few studies have compared these techniques in order to establish the best method. We will compare an older technique using a metal handle and blade that allows for direct visualization of the vocal cords (direct laryngoscopy) to a newer technique that employs a fiberoptic bundle imbedded in a handle that allows indirect visualization of the vocal cords during placement of the artificial airway. The newer technique has the theoretical advantage of being more useful in patients with abnormal airways which are frequently encountered in trauma patients. Since both techniques are currently employed routinely in our institution, we will randomize all trauma admission to have an initial attempt with one of the two techniques in order to perform a randomized, unblinded trial.

ELIGIBILITY:
Inclusion Criteria:

* require emergency intubation

Exclusion Criteria:

* age < 18
* require surgical airway on initial assessment
* have known or strongly suspected spinal cord injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 623 (Actual)
Dates: Start 2008-07; Primary Completion 2016-11-16 (Actual); Study Completion 2016-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dale Yeatts, MD, Principal Investigator — University of Maryland
Locations (1):
- R Adams Cowley Shock Trauma Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
None exists

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Direct Laryngoscope | Video Laryngoscope
Started | 320 | 303
Completed | 320 | 303
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Direct Laryngoscope | Video Laryngoscope | Total
Number analyzed (Participants) | 320 | 303 | 623
Age, Continuous [Mean (Full Range); unit: years] | 43 [18 to 65] | 42 [18 to 65] | 43 [18 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 87 | 163
  Male | 244 | 216 | 460
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 320 | 303 | 623

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Survived to Hospital Discharge
Description: Assessment of whether or not the patient was discharged alive from the study center
Time Frame: 2 weeks, on average
Measure: Count of Participants; unit: Participants
Arm/Group | Direct Laryngoscope | Video Laryngoscope
Number analyzed (Participants) | 320 | 303
Participants | 296 | 275

2. Secondary Outcome: Length of Time to Perform the Intubation Procedure
Description: How long (seconds) it takes the provider to perform the intubation procedure.
Time Frame: Up to 100 seconds
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Direct Laryngoscope | Video Laryngoscope
Number analyzed (Participants) | 296 | 275
seconds | 40 [24 to 68] | 56 [40 to 81]

ADVERSE EVENTS:
Arm/Group | Direct Laryngoscope | Video Laryngoscope
Serious Adverse Events (participants affected / at risk) | 0/320 | 0/303
Other Adverse Events (participants affected / at risk) | 0/320 | 0/303

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes